CLINICAL TRIAL: NCT00151034
Title: Phase II Evaluation of Trastuzumab (Herceptin), Paclitaxel, Carboplatin, and Gemcitabine in the Treatment of Advanced Urothelial Cancer
Brief Title: Trastuzumab (Herceptin), Paclitaxel, Carboplatin and Gemcitabine in Advanced Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 9955
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Urologic Neoplasms
Keywords: Urothelial Cancer; Herceptin; Advanced Urothelial Cancer
MeSH Terms: conditions — Urologic Neoplasms | interventions — Trastuzumab; Paclitaxel; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Herceptin (Experimental): Herceptin - 4mg/kg day 1 of cycle 1; 2mg/kg day 8 and 15 of cycle 1 and subsequent cycles.
  Paclitaxel - 200mg/m^2 on day 1 Carboplatin - AUC 5 on day 1 Gemcitabine - 800 mg/m^2 on day 1 and 8
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Trastuzumab
  Other Names: Herceptin
Drug: Paclitaxel
Drug: Carboplatin
Drug: Gemcitabine

SUMMARY:
Purpose: The purpose of this study is to evaluate the efficacy and safety of treatment with trastuzumab (Herceptin) along with the three other chemotherapy drugs, paclitaxel, carboplatin and gemcitabine, in patients who have advanced urothelial cancer. This clinical trial will also collect information (alternative therapy, response rates, overall survival) from enrolled patients with HER2 negative tumors who are ineligible to receive study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of urothelial carcinoma (TCC or Squamous) that is either metastatic or locally recurrent and not curable by surgery or radiation therapy.
* All patients must have tissue from either the primary or metastatic site tested for HER2 status determination. Patients with Her-2 negative tumors are not eligible for treatment on this protocol.
* All patients must have a blood sample drawn for HER2 serologic testing.
* If the available tissue is from the primary tumor and is HER2 negative and if the serum is negative, to qualify for the study a biopsy of a metastatic site should be done and the patient will be eligible ONLY if this demonstrates HER2 over-expression.
* Patients may not have received prior systemic chemotherapy for metastatic disease. Patients may have received adjuvant chemotherapy if completed at least 6 months prior to beginning this protocol treatment.
* Patients may not have cardiac disease and must have adequate cardiac function (ejection fraction > 50% or higher than the lower limit of institutional normal) as determined by a MUGA scan or 2-D echocardiogram within 4 weeks from registration, and no evidence of symptomatic coronary artery disease (baseline EKG must show no active ischemia). Patients must not have history of congestive heart failure.
* If patients have received prior radiation therapy, disease must be present outside of radiated fields and at least 4 weeks must have elapsed since discontinuation of that therapy.

Exclusion Criteria:

* Pregnant or lactating women may not participate.
* HIV - positive patients may not participate. This is to avoid additional complications that immune suppression and HIV infection may cause due to the intense nature of the chemotherapy in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2000-09; Primary Completion 2004-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The Number of Toxicities Experienced by Treated Patients | 30 Days Post Treatment
  The primary objective of the study is to evaluate the toxicity profile of combination of herceptin, paclitaxel, carboplatin and gemcitabine in patients with locally recurrent or metastatic urothelial carcinoma who overexpress HER2.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hussain, MD, Principal Investigator — The University of Michigan Comprehensive Cancer Center
Locations (11):
- United States (11):
  - California City of Hope National Medical Group, Duarte, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - U.C. Davis Medical Center, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania